CLINICAL TRIAL: NCT02927756
Title: Italian Multicenter Retrospective Observational Study on Transformed Lymphomas
Acronym: FLT-Oss-2015
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Barbara Botto, MD, A.O.U. Città della Salute e della Scienza
Other Study IDs: FLT-Oss-2015
Record Dates: First submitted 2016-09-28; First posted 2016-10-07 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Non-Hodgkin Lymphoma Transformed Recurrent
Keywords: Non-Hodgkin Lymphoma Transformed Recurrent; Discordant Lymphomas; Composite Lymphomas; Follicular Lymphoma; Aggressive Lymphoma
MeSH Terms: conditions — Composite Lymphoma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study purpose is to evaluate treatment outcome and survival in patient with aggressive lymphomas transformed from Follicular Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed transformed Follicular Lymphoma
* Age > 18 years
* Histological transformation between January 2002 and December 2014
* Availability of data about treatment and outcome

Exclusion Criteria:

* Other lymphoma diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with histologically confirmed diagnosis of Transformed Follicular Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From first response to last follow-up for at least 2 years (up to 15 years)
  Time from last response to nearest relapse or follow-up
Overall Survival | Date of last follow-up for at least 2 years (up to 15 years)
  Time to last follow-up or death

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Botto, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- SC Ematologia - AOU Città della Salute e della Scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: Yes
paper publication